CLINICAL TRIAL: NCT03682562
Title: Diagnostic Accuracy of Salivary DNA Integrity Index in Oral Malignant and Premalignant Lesions
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Adel Azab, Researcher, Cairo University
Other Study IDs: N1P1H1D1
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Oral Cancer; Oral Lichen Planus; Oral Leukoplakia
MeSH Terms: conditions — Mouth Neoplasms; Lichen Planus, Oral; Leukoplakia, Oral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Salivary Samples will be obtained for DNA extraction, Biosamples will be stored in -80 degrees after patient's consent
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oral Cancer: Patients diagnosed clinically and histopathologically as having oral cancer.
  Interventions: Diagnostic Test: DNA Integrity Index
- Premalignant Oral Lesions: Patients diagnosed clinically and histopathologically with either leukoplakia or oral lichen planus as stated by modified WHO criteria
  Interventions: Diagnostic Test: DNA Integrity Index
- Normal Subjects: Patients who give a history of:
  * No smoking
  * No alcohol
  * No systemic disease; and who on conventional oral examination have:
  * No visible oral lesions on conventional oral examination .
  * Good oral hygiene.
  Interventions: Diagnostic Test: DNA Integrity Index

INTERVENTIONS:
Diagnostic Test: DNA Integrity Index — This test will be performed for ALL three groups:
  Sample collection:
  Patients will be given a sterile cup containing 5mL saline solution with which they will vigorously rinse their mouth while rubbing their tongues against the oral mucosa for 30 seconds, then spit it back into the cup. The solution will then be used for DNA extraction.
  DNA integrity analysis:
  The DNA integrity will be done through measuring a housekeeping gene using competitive polymerase chain reaction where the isolated DNA will be combined with DNA capture probes for sequence-specific DNA fragments. The DNA integrity index will be calculated as the ratio of the concentration of longer DNA fragments to the ratio of shorter ones.

SUMMARY:
This study aims to identify the accuracy of DNA integrity index in differentiating between oral premalignant lesions and oral cancer.

DETAILED DESCRIPTION:
As stated by the U.S. Preventive Services Task Force and the National Institute of Dental and Craniofacial Research, the main screening test for oral cancer remains conventional oral examination of the oral cavity. Most cases of oral cancer are preceded by a clinically visible lesion. These lesions are called oral potentially malignant disorders. These are leukoplakia, erythroplakia, oral submucous fibrosis, oral lichen planus and discoid lupus erythematosis. Leukoplakia has a reported annual transformation rate of 2-3%, while OLP has a rate of 0.5% .

Full thickness tissue biopsy is the "gold standard" for diagnosing suspicious lesions should they be encountered during COE. However, oral biopsy is an invasive technique that can be challenging in sites as the floor of the mouth or the soft palate . The invasive nature of a biopsy also makes it unsuitable for cancer screening in high-risk populations.

Thus there is a need for a diagnostic aid that can help primary care providers determine which patients need to be biopsied or referred to a specialist.

Nucleic acids can be released actively or passively into the circulation by both living and dead cells, where the latter is considered the predominant source. Programmed cell death gives neatly digested DNA fragments of approximately 180 bp in length. In case of solid tumors, cell-free DNA is released through necrosis which generates longer DNA fragments due to haphazard and incomplete digestion of DNA. Thus, the integrity of the DNA fragment can determine its origin making DNA integrity a potential marker for oral cancer.

The DNA integrity index (DII) is the ratio between the longer DNA fragments to the shorter ones. A higher index has been reported in breast, prostate, liver and cervical cancer. Jiang et al. 2006 found that the DNA integrity index was significantly higher in oral cancer patients than in normal ones and reported a sensitivity and specificity values of 84.5% 83% respectively . The next step for such a marker would be early quantification of performance in clinical settings to determine if it is possible to extrapolate cut off values.

ELIGIBILITY:
Patients in this study will be divided into three groups:

Group I: Patients diagnosed histopathologically with oral cancer recruited from the National Cancer Institute, who have yet to receive treatment.

Group II: Healthy Controls

Inclusion Criteria:

* No visible oral lesions as detected by conventional oral examination
* Good oral hygiene, with healthy gingival tissues
* Non-smokers
* No systemic disease Group III: Patients diagnosed with oral lichen planus according to the modified WHO (van der Meij and van der Waal, 2003)diagnostic criteria not receiving treatment at least 8 weeks prior to enrollment.

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Group I: (Clinical examination and Biopsy) Patients diagnosed clinically and histopathologically as having oral cancer. Group II: (History and Clinical examination)
  Patients who give a history of:
  * No smoking
  * No alcohol
  * No systemic disease; and who on conventional oral examination(National Institute of Dental and Craniofacial Research, 2013b) have:
  * No visible oral lesions on conventional oral examination .
  * Good oral hygiene. Group III: (Clinical examination and Biopsy) Patients diagnosed clinically and histopathologically with oral lichen planus as stated by modified WHO criteria (van der Meij and van der Waal, 2003).
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Difference in DNA Integrity Index | 1 month after the end of patient recruitment
  The DNA integrity will be compared between the three group to determine whether there is a difference between them in that aspect or not

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
According to the mode of data entry, if it is solely numerical it can be more easily shared and deposited on repositories, however patient clinical photos may not be possible to share